CLINICAL TRIAL: NCT01330628
Title: EXCImer Laser Randomized Controlled Study for Treatment of FemoropopliTEal In-Stent Restenosis
Brief Title: Randomized Study of Laser and Balloon Angioplasty Versus Balloon Angioplasty to Treat Peripheral In-stent Restenosis
Acronym: EXCITE ISR
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D013474
Record Dates: First submitted 2011-04-04; First posted 2011-04-07 (Estimated); Results first posted 2016-06-15 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-07

CONDITIONS: Peripheral Arterial Disease
Keywords: peripheral arterial disease; in stent restenosis; peripheral vascular disease
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Vascular Diseases | interventions — Angioplasty, Balloon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laser atherectomy and PTA (Experimental): laser, then balloon angioplasty
  Interventions: Device: Turbo Elite Laser and Turbo Tandem Laser Guide Catheters
- Balloon angioplasty (Active Comparator)
  Interventions: Procedure: Balloon angioplasty

INTERVENTIONS:
Device: Turbo Elite Laser and Turbo Tandem Laser Guide Catheters — application of laser energy to remove blockage followed by standard balloon angioplasty
  Arms: Laser atherectomy and PTA
Procedure: Balloon angioplasty — standard balloon catheters for PTA
  Arms: Balloon angioplasty

SUMMARY:
The purpose of the study is to evaluate the safety and efficacy of laser atherectomy with balloon angioplasty compared to balloon angioplasty alone in the treatment of above the knee peripheral artery in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

* PAD with Rutherford class 1-4
* Resting ABI <0.9 or abnormal exercise ABI <0.9
* History of previous femoropopliteal nitinol stenting
* Angiographic significant restenosis (>=50%)
* Target lesion length >=4 cm; no more than 3 cm outside stent at either end
* Vessel diameter >=5 mm and <=7 mm
* At least one widely patent tibial or peroneal artery to the foot

Exclusion Criteria:

* Patient is pregnant or breast feeding
* Evidence of acute limb ischemia
* Life expectancy <12 months
* CVA within 60 days of screening
* Myocardial infarction within 60 days of procedure
* Known allergy to contract media
* Known contraindication to aspirin, antiplatelet and anti-coagulation therapies
* Uncontrolled hypercoagulability
* Present or suspected systemic infection in target limb
* Serum creatinine >= 2.5 mg/dl unless dialysis dependent
* Previous treatment to target vessel within 3 months of study procedure
* Drug eluting stents or covered stents in target lesion
* Ipsilateral and/or contralateral iliac stenosis >= 50% DS that is not successfully treated prior to index procedure or with final residual stenosis <= 30% documented by angiography
* Planned or predicted cardiovascular surgical or interventional procedures prior to completion of the 30-day follow-up
* Identification of any lesion below the target stent in the treated leg >50% that will require preplanned or predicted treatment within 30 days(prior to the 6 month follow up)
* Tibial artery containing a >50% Diameter Stenosis (DS) by visual estimate after popliteal
* Grade 4 or 5 stent fracture affecting target stent or proximal to the target stent, or where evidence of stent protrusion into the lumen is noted on angiography in 2 orthogonal views.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2011-06; Primary Completion 2014-03 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Dippel, MD, Principal Investigator — Genesis Health System
Locations (34):
- United States (33):
  - St. Vincent's East, Birmingham, Alabama
  - Thomas Hospital, Fairhope, Alabama
  - St. Vincent Heart Clinic Arkansas, Little Rock, Arkansas
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - UC-Davis Medical Centers, Sacramento, California
  - Yale - New Haven Hospital, New Haven, Connecticut
  - Washington Hospital Center, Washington D.C., District of Columbia
  - The Cardiac and Vascular Institute, Gainesville, Florida
  - Memorial Regional Hospital, Hollywood, Florida
  - Mount Sinai Medical Center, Miami, Florida
  - St. John's Hospital, Springfield, Illinois
  - Community Hospital, Munster, Indiana
  - Genesis Health System, Davenport, Iowa
  - Cardiovascular Consultants, Bossier City, Louisiana
  - Regional Medical center of Acadiana, Lafayette, Louisiana
  - Opelousas General Hospital, Opelousas, Louisiana
  - Steward - St. Elizabeth's, Boston, Massachusetts
  - St. John's - Providence Hospital, Southfield, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Deborah Heart and Lung, Browns Mills, New Jersey
  - New York University, New York, New York
  - Coastal Surgery Specialists, Wilmington, North Carolina
  - Bryn Mawr, Bryn Mawr, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Wellmont Holston Valley Medical, Kingsport, Tennessee
  - Presbyterian Hospital of Dallas, Dallas, Texas
  - El Paso Cardiac and Endovascular Center, El Paso, Texas
  - Tyler Cardiac and Endovascular Center, Tyler, Texas
  - Providence Health Center, Waco, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Wheaton Franciscan Healthcare - All Saints Hospital, Milwaukee, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
- Transcatheter Medical Inc., San Juan, Puerto Rico

REFERENCES:
- [Derived] Dippel EJ, Makam P, Kovach R, George JC, Patlola R, Metzger DC, Mena-Hurtado C, Beasley R, Soukas P, Colon-Hernandez PJ, Stark MA, Walker C; EXCITE ISR Investigators. Randomized controlled study of excimer laser atherectomy for treatment of femoropopliteal in-stent restenosis: initial results from the EXCITE ISR trial (EXCImer Laser Randomized Controlled Study for Treatment of FemoropopliTEal In-Stent Restenosis). JACC Cardiovasc Interv. 2015 Jan;8(1 Pt A):92-101. doi: 10.1016/j.jcin.2014.09.009. Epub 2014 Dec 10. PMID 25499305

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Laser Atherectomy and PTA | Balloon Angioplasty
Started | 170 | 82
30 Day Follow-up | 165 | 73
6 Month Follow-up | 135 | 60
Completed | 100 | 42
Not Completed | 70 | 40
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 5 | 6
Not completed — Adverse Event | 44 | 25
Not completed — Withdrawn | 18 | 6
Not completed — Didn't receive study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Laser Atherectomy and PTA | Balloon Angioplasty | Total
Number analyzed (Participants) | 170 | 82 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.6 (9.8) | 67.9 (10.3) | 68.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 31 | 95
  Male | 106 | 51 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 12 | 33
  Not Hispanic or Latino | 149 | 70 | 219
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 22 | 8 | 30
  White | 144 | 74 | 218
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 170 | 82 | 252

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Target Lesion Revascularization (TLR)
Description: Number of participants free from Target Lesion Revascularization (TLR) through 6 months follow-up.
Time Frame: 6 months
Population: The number of participants analyzed for this endpoint does not match with the Participant Flow 6 Month Follow-up population. A subject may not complete a 6 Month Follow-up due to missing the visit, being lost to follow-up, etc., but if they had a TLR prior to this time point, they would still be included in this outcome analysis.
Measure: Number; unit: # of participants free from TLR
Arm/Group | Laser Atherectomy and PTA | Balloon Angioplasty
Number analyzed (Participants) | 157 | 73
# of participants free from TLR | 123 | 43

2. Primary Outcome: Freedom From Major Adverse Events (MAE)
Description: Number of participants free from Major Adverse Events (MAE) at 30 days. MAE are defined all cause death, major amputation in the target limb, or target lesion revascularization (TLR) from procedure to 30 days (±7 days).
Time Frame: 30 days
Population: The number of participants analyzed for this endpoint does not match with the Participant Flow 30 Day Follow-up population. If a subject did not complete a 30 Day Follow-up due to missing the visit or lost to follow-up, but had an MAE prior to this time point, they would still be included in this outcome analysis.
Measure: Number; unit: # of participants free from MAE
Arm/Group | Laser Atherectomy and PTA | Balloon Angioplasty
Number analyzed (Participants) | 167 | 77
# of participants free from MAE | 158 | 61

ADVERSE EVENTS:
Time Frame: Through 1 year
Description: Specific study related terms (death, amputation and/or TLR) are in the Primary Outcomes Table. To summarize the remaining events, they were categorized into general organ class. The general organ classes are inclusive of the specific study related events. All events were adjudicated and categorized by an independent Clinical Events Committee.
Arm/Group | Laser Atherectomy and PTA | Balloon Angioplasty
Serious Adverse Events (participants affected / at risk) | 117/170 | 56/82
Other Adverse Events (participants affected / at risk) | 88/170 | 34/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Atherectomy and PTA (N=170) | Balloon Angioplasty (N=82)
Infection SAEs (Infections and infestations) | 3 | 4
Cardiac SAEs (Cardiac disorders) | 19 | 8
Other SAEs (General disorders) | 25 | 12
Gastrointestinal SAEs (Gastrointestinal disorders) | 9 | 6
Neurological SAEs (Nervous system disorders) | 4 | 5
Blood related disorder SAEs (Blood and lymphatic system disorders) | 5 | 1
Vascular SAEs (Vascular disorders) | 96 | 48
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Atherectomy and PTA (N=170) | Balloon Angioplasty (N=82)
Infection (Infections and infestations) | 9 | 4
Cardiac (Cardiac disorders) | 15 | 4
Other AEs (General disorders) | 40 | 8
Gastrointestinal (Gastrointestinal disorders) | 10 | 3
Neurological (Nervous system disorders) | 8 | 3
Blood related disorders (Blood and lymphatic system disorders) | 7 | 5
Vascular (Vascular disorders) | 53 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less